CLINICAL TRIAL: NCT06433791
Title: Phase 1, Single-Center, Dose-Escalating, Open-Label, Safety Clinical Trial of Parenteral Ascorbate-Meglumine As a Novel Magnetic Resonance Imaging (MRI)-guided Adjunctive Therapeutic for Stereotactic Radiosurgery (SRS)
Brief Title: Evaluation of Ascorbate-Meglumine Therapeutic for SRS
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: LadeRx LLC (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LadeRX; NCT03927625 (obsolete NCT alias)
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Safety
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ascorbate Meglumine dose 1 (Experimental): Patients receiving Stereotactic Radiosurgery (SRS) treatment for cancer metastatic to the brain from an extracranial primary site with a contrast-enhanced Magnetic Resonance Imaging (MR) scan showing 1-3 brain metastases, including post-operative patients with 1-3 residual metastases. The first cohort of patients will receive ascorbate-meglumine at a dose administration rate of 0.16 g/min for 60 minutes.
  Interventions:
  Drug: Ascorbate-Meglumine
  Interventions: Drug: Ascorbate-Meglumine
- Ascorbate Meglumine dose 2 (Experimental): Patients receiving SRS treatment for cancer metastatic to the brain from an extracranial primary site with a contrast-enhanced MRI scan showing 1-3 brain metastases, including post-operative patients with 1-3 residual metastases.The second cohort of patients will receive ascorbate-meglumine at a dose administration rate of 0.31 g/min for 60 minutes.
  Interventions:
  Drug: Ascorbate-Meglumine
  Interventions: Drug: Ascorbate-Meglumine
- Ascorbate Meglumine dose 3 (Experimental): Patients receiving SRS treatment for cancer metastatic to the brain from an extracranial primary site with a contrast-enhanced MRI scan showing 1-3 brain metastases, includingpost-operative patients with 1-3 residual metastases. The third cohort of patients will receive ascorbate-meglumine at a dose administration rate of 0.63 g/min for 60 minutes.
  Interventions:
  Drug: Ascorbate-Meglumine
  Interventions: Drug: Ascorbate-Meglumine
- Ascorbate Meglumine dose 4 (Experimental): Patients receiving SRS treatment for cancer metastatic to the brain from an extracranial primary site with a contrast-enhanced MRI scan showing 1-3 brain metastases, includingpost-operative patients with 1-3 residual metastases. The fourth cohort of patients will receive ascorbate-meglumine at a dose administration rate of 1.25 g/min for 60 minutes.
  Interventions:
  Drug: Ascorbate-Meglumine
  Interventions: Drug: Ascorbate-Meglumine

INTERVENTIONS:
Drug: Ascorbate-Meglumine — Ascorbate, meglumine and sodium salt made by combining 375 mM sodium ascorbate,125 mM ascorbic acid and 125 mM meglumine in sterile water for injection
  Other Names: Vitamin C

SUMMARY:
Phase 1, Single-Center, Dose-Escalating, Open-Label, Safety Clinical Trial of Parenteral Ascorbate-Meglumine as a Novel Magnetic Resonance Imaging (MRI)-guided Adjunctive Therapeutic for Stereotactic Radiosurgery (SRS)

DETAILED DESCRIPTION:
Phase 1, single-center, open-label study in subjects receiving Stereotactic Radiosurgery (SRS) for brain metastases. The study will consist of 4 principal cohorts (n=3 in each cohort). Each cohort will receive an escalating dose of ascorbate-meglumine as an Magnetic Resonance Imaging (MRI)-detectable adjunctive therapeutic to SRS.

Subjects will complete a planning MRI for SRS with gadolinium- diethylenetriamine penta-acetic acid (GD-DPTA) per standard of care for SRS. Forty-eight hours after the planning MRI, the subjects will complete the study MRI with ascorbate-meglumine contrast agent. Each cohort will receive an escalating dose of ascorbate-meglumine by intravenous administration over 1 hour during the MRI. The total dose of ascorbate-meglumine will escalate from the first cohort to the next cohort in a sequential manner. During ascorbate-meglumine infusion, MRI scans will be performed to evaluate the contrast effect and PK blood draws will occur at defined time points.

Patients will return for the SRS procedure within 1 week following the planning MRI per standard of care. During SRS, subjects will receive a second dose of ascorbate-meglumine as an adjunctive therapeutic.

Patients will enter into a follow up phase within 2 weeks after the SRS procedure per standard of care.

The primary endpoint is to evaluate the safety of parenteral ascorbate-meglumine as a MRI-detectable adjunctive therapeutic to SRS.

ELIGIBILITY:
Inclusion Criteria:

* Primary cancer diagnosis with newly diagnosed brain metastases
* Diagnostic MRI demonstrates the presence of 1 to 3 intact (not previously irradiated or resected) brain metastases.
* Maximum tumor diameter ≤ 2.5 cm for the largest lesion determined during the planning MRI
* Plan of care must include Stereotactic Radiosurgery (SRS)
* SRS treatment plan must be delivered as a single RT fraction
* Age 18 years and older
* Life expectancy of at least 3 months
* GPA score 0.5 or greater
* Capable of providing written informed consent to participate in the study

Exclusion Criteria:

* Primary lesion with radiosensitive histology (i.e., small cell carcinoma, germ-cell tumors, lymphoma, leukemia, and multiple myeloma)
* Metastases in the brain stem, pons or medulla or within 3 mm of the optic apparatus (such that some portion of the optic nerve or chiasm would receive a radiation dose > 10 Gy SRS in one single fraction)
* Previous whole-brain radiation (previous SRS to or resection of other brain lesions is permitted if more than 3 months prior to the date of enrollment on this protocol)
* Pregnancy
* History or manifestation of glucose-6-phosphate dehydrogenase (G6PD) enzyme deficiency
* History of oxalate kidney stones
* History of iron overload or hemochromatosis
* History of allergy to ascorbic acid
* Anuria, dehydration, serum albumin <3.0 g/dL, severe pulmonary congestion or pulmonary edema or fixed low cardiac input since all are conditions for which osmotic diuresis are contraindicated .
* Subjects who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide.
* Subjects who are on strong inducers, inhibitors or substrates of CYP within 3 days of planned administration of study ascorbate-meglumine.
* Subjects for which MRI is contra-indicated (for example a pacemaker/recent surgery with orthopedic prosthesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-05-17 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by adverse events | 1 week after receiving study drug with SRS
  Adverse events will be monitored in patients receiving ascorbate-meglumine during Stereotactic Radiosurgery (SRS)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkpatrick, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No